CLINICAL TRIAL: NCT01983462
Title: Vascular Dysfunction in Human Obesity Hypertension: Integrative Role of Sympathetic and Renin-Angiotensin Systems
Brief Title: Vascular Dysfunction in Human Obesity Hypertension
Acronym: VANISH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding expired
Sponsor: Gary L. Pierce (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Gary L. Pierce, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201307779
Record Dates: First submitted 2013-10-30; First posted 2013-11-14 (Estimated); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Prehypertension; Hypertension
Keywords: Prehypertension; Hypertension; Obese; Sympathetic Nervous System; renin-angiotensin system; Endothelial function
MeSH Terms: conditions — Obesity; Prehypertension; Hypertension | interventions — Clonidine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clonidine (Experimental): Oral 0.2 mg/day (0.1 mg bid)for 4 weeks
  Interventions: Drug: Clonidine
- Hydrochlorothiazide (Active Comparator): Oral, 12.5 mg/day qd, 4 weeks
  Interventions: Drug: Hydrochlorothiazide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine
  Other Names: Catapress
  Arms: Clonidine
Drug: Hydrochlorothiazide
  Arms: Hydrochlorothiazide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to test the effects of blocking sympathetic nerve activity with a drug called clonidine on blood vessel function and muscle nerve activity in adults who are obese and have high blood pressure.

The cohort of subjects will consist of 69 healthy young men and women age 18-79 years who are obese, defined as a body mass index > or = to 30 kg/m2, who have untreated systolic hypertension (systolic blood pressure > or = to 130 - <180 mmHg- average of at least 3 measurements 2 min apart after 10 min seated resting position). These 69 subjects will then be randomized to 3 treatment arms: clonidine (0.1 mg/day), hydrochlorothiazide (25 mg/day) or placebo for 4 weeks in years 1 and 2. All tablets will be encapsulated by to look identical. Subjects will randomly (1:1:1) receive one of the following combinations in a double-blind, placebo-controlled design:

1. Oral clonidine (0.1 mg twice/day)
2. Oral hydrochlorothiazide (12.5 mg twice/day)
3. Oral placebo

I

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Systolic blood pressure >/= 130 mmHg and <180 mmHg
* Age is > or = 18 and < or = 79 years of age
* Weight stable (+/- 5 lbs) for the previous 3 months
* Healthy, as determined by health history questionnaire, blood chemistries, 12-lead ECG
* Blood chemistries indicative of normal renal (creatinine <2.0 mg/dl), liver (<3 times upper limit for ALT, AST), and thyroid function (TSH between 0.4 - 5.0 mU/L)
* If currently receiving treatment with or taking any of the following supplements, be willing and able to discontinue taking them for 2 weeks prior and throughout the treatment period: Vitamin C, E or other multivitamins containing vitamin C or E; or omega-3 fatty acids.
* No history of cardiovascular disease (e.g., heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy), Type 1 or Type 2 diabetes, or peripheral arterial disease
* Non-smokers, defined as no history of smoking or no smoking for at least the past 1 year
* Normal resting 12-lead ECG (no evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter)

Exclusion Criteria:

* Systolic blood pressure >/=180 mmHg or diastolic blood pressure >110 mmHg
* History of cardiovascular disease such as heart angioplasty/stent or bypass surgery, myocardial infarction, stroke, heart failure with or without left ventricular ejection fraction <40%, cardiomyopathy, valvular heart disease, cardiomyopathy, heart transplantation, Type 2 and Type 1 diabetes
* Smoking or history of smoking within past one year
* History of gastric ulcers, bleeding disorders, dyspepsia, severe gastroesophageal reflux disease (GERD), or metabolic acidosis
* History of chronic obstructive pulmonary disease (COPD)
* Abnormal resting 12-lead ECG (e.g., evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter)
* Serious neurologic disorders including seizures
* History of renal failure, dialysis or kidney transplant
* Serum creatinine > 2.0 mg/dL, or hepatic enzyme (ALT/AST) concentrations > 3 times the upper limit of normal
* History of HIV infection, hepatic cirrhosis, other preexisting liver disease, or positive HIV, Hepatitis B or C test at screening.
* Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* History of recent chicken pox, shingles or influenza (ie., risk of Reye's syndrome)
* Recent flu-like symptoms within the past 2 weeks
* Pregnant or breastfeeding at screening, or planning to become pregnant (self or partner) at any time during the study. A urinary pregnancy test will be done on all females. If test is positive, the subject will be excluded.
* Women with history of hormone replacement therapy within the past 6 months
* History of rheumatoid arthritis, Grave's disease, systemic lupus erythematosis, and Wegener's granulomatosis;
* Taking lipid lowering (e.g., statins, niacin), glycemic control (e.g. metformin, insulin), anticoagulation, anti-seizure, anti-depression or antipsychotic agents
* History of co-morbid condition that would limit life expectancy to < 6 months.
* Taking chronic non-steroidal anti-inflammatory drugs (NSAIDS) such as aspirin, indomethacin, naproxen, acetaminophen (Tylenol), ibuprofen (Advil, Motrin) and not able or willing to go off of for 2 weeks prior and during the study
* Taking cox-2 inhibitors (Celebrex, Vioxx, etc) or allopurinol (Zyloprim, Lopurin, Allopurin)
* Taking blood thinners such as coumadin (Warfarin), enoxaparin (Lovenox); clopidogrel (Plavix); dipyridamole (Persantine); heparin;
* Taking diabetic medications (Metformin, glyburide, insulin, etc.), thiazolidinediones (Avandia, Rezulin, Actos);
* Taking steroids or biologics : corticosteroids (prednisone); methotrexate, infliximab (Remicade), etanercept (Enbrel); anakinra;
* Taking thyroid medications such as levothyroxine (Levoxyl, Synthroid, Levoxyl, Unithroid); Levodopa;
* Taking Phosphodiesterase (PDE) 5 inhibitors (e.g., Viagra®, Cialis®, Levitra®, or Revatio®); PDE 3 inhibitors (e.g., cilostazol, milrinone, or vesnarinone); lithium
* May participate if no use of the following medications in the 48 hours prior to experimental visits: naproxen (Aleve), acetaminophen (Tylenol), ibuprofen (Advil, Motrin), other any non-steroidal anti-inflammatory drugs (NSAIDS)
* Vulnerable populations (prisoners, etc.)
* Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
* History of alcohol abuse or >10 alcoholic units per week (1 unit= 1 beer, 1 glass of wine, 1 mixed cocktail containing 1 oz alcohol)
* On weight loss drugs (e.g., Xenical (orlistat), Meridia (sibutramine), Acutrim (phenylpropanol-amine), or similar over-the-counter medications) within 3 months of screening
* Any surgery within 30 days of screening

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Pierce, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized to clonidine, HCTZ or placebo for 4 weeks
Groups:
- Clonidine: Oral 0.2 mg/day (0.1 mg bid)for 4 weeks
  Clonidine
- Hydrochlorothiazide: Oral, 12.5 mg/day qd, 4 weeks
  Hydrochlorothiazide
Period: Overall Study
Arm/Group | Clonidine | Hydrochlorothiazide | Placebo
Started | 11 | 11 | 11
Completed | 10 | 11 | 11
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine | Hydrochlorothiazide | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 11 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 10 | 31
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (18) | 31 (10) | 37 (19) | 35 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 8
  Male | 9 | 10 | 6 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 10 | 11 | 10 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 5
  White | 6 | 6 | 10 | 22
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Aortic Stiffness
Description: Carotid-femoral pulse wave velocity (PWV)
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: meters/sec
Arm/Group | Clonidine | Hydrochlorothiazide | Placebo
Number analyzed (Participants) | 10 | 11 | 11
meters/sec
  Baseline | 7.9 (0.7) | 7.0 (0.4) | 8.1 (1.0)
  4 weeks | 7.3 (0.6) | 7.0 (0.3) | 8.0 (1.2)

2. Secondary Outcome: 24 Hour Average Systolic Blood Pressure
Description: 24 hour ambulatory systolic blood pressure
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Clonidine | Hydrochlorothiazide | Placebo
Number analyzed (Participants) | 10 | 11 | 9
mmHg
  Baseline | 133 (3) | 135 (2) | 133 (2)
  4 weeks | 126 (3) | 131 (2) | 134 (2)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Clonidine | Hydrochlorothiazide | Placebo
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 0/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine (N=10) | Hydrochlorothiazide (N=11) | Placebo (N=11)
Mild hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT01983462/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT01983462/SAP_001.pdf